CLINICAL TRIAL: NCT04610463
Title: Evaluation of the Severity of Right to Left Shunt in Patent Foraneb Ovale Patients After Systemic Embolism
Brief Title: Evaluation of the Severity of Right to Left Shunt in PFO Patients After Systemic Embolism
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University Hospital Hradec Kralove (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: MEASURE-PFO
Record Dates: First submitted 2020-06-12; First posted 2020-10-30 (Actual); Last update posted 2020-10-30 (Actual); Status verified 2020-10

CONDITIONS: Patent Foramen Ovale; Embolism
Keywords: Patent foramen ovale; Systemic Embolism; Cardiac Shunt; Right to left shunt; Hemodynamics
MeSH Terms: conditions — Foramen Ovale, Patent; Embolism

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Standard (Other): Subjects indicated for patent foramen ovale closure to prevent a relapse of systemic embolism
  Interventions: Diagnostic Test: Cardiac flow measurement

INTERVENTIONS:
Diagnostic Test: Cardiac flow measurement — Catheterized hemodynamics evaluation - a measurement of systemic flow and pulmonary flow, R-L shunt, L-R shunt using the INNTHERM® system, prior to PFO closure using a common PFO-occluder (within one catheterization intervention).

SUMMARY:
The aim of the project is to identify new risk indicators of PFO. The evaluation of the R-L shunt is based on the newly developed precise measurement technique. Moreover, this measurement of R-L shunt is feasible in a case when R-L shunt is present only intermittently. Multicentric study with 150 patients.

DETAILED DESCRIPTION:
The aim of the proposed project is to identify new risk indicators of PFO. The evaluation of the R-L shunt is based on the newly developed precise measurement technique. Moreover, this measurement of R-L shunt is feasible in a case when R-L shunt is present only intermittently.

Detection and quantification of R-L shunt will be realized by the original INNTHERM® ® system (Innova Medical s.r.o., Velká Dobrá). This system is based on the principle of thermodilution.

The basic assumption of our study is the hypothesis, that the size of the R-L shunt (and especially its maximum size during intra-abdominal pressure increase) is a risk factor for the development of paradoxical embolism (from pulmonary to systemic circulation). The most critical consequence of paradoxical embolism is the development of ischemic stroke.

Such measurement with an unequivocal accuracy has never been done so far, due a lack of technology precise enough.

Precise quantification of R-L shunt will allow a more accurate prediction of high-risk patients, especially after correlation with commonly used methods. PFO is now an indication for implantation of percutaneous occlusion device only in case of secondary prevention of stroke, i.e. in a group of patients who have had an ischemic stroke.

Prospectively, precise and better identification of a risk group of these patients could lead to cost reduction of treatment. This cost reduction is crucial for young working-age patients who can be treated before a major irreversible brain injury occurs.

A parameter applicable in primary prevention saves the cost of ischemic stroke treatment and other systemic embolism; additionally it will contribute to cost reduction during aftercare treatment.

ELIGIBILITY:
Inclusion Criteria:

1. Male and female patients aged ≥18 and < 60 years
2. Cryptogenic stroke or Systemic embolization due to paradoxical embolization via Patent Foramen Ovale
3. The patient indicated for occlusion of PFO with catheter occluder

Exclusion Criteria:

1. Inability to perform spiroergometry
2. Inability to perform Transesophageal echocardiography (TEE)
3. Inability to perform proper Valsalva maneuver
4. Inability to understand and/or signed informed consent form
5. Contraindication of Patent Foramen Ovale occlusion by any medical reason or patient refusal

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 150 (Estimated)
Dates: Start 2020-09-25 (Actual); Primary Completion 2023-12 (Estimated); Study Completion 2023-12 (Estimated)

PRIMARY OUTCOMES:
Quantification of R-L shunt namely | Up to 24 weeks
  Right-to Left shunt will be measured and quantified using by the novel system for measurement of Cardiac flow- Inntherm. We will obtain these hemodynamics parameters: Systemic blood flow (SBF) pulmonary blood (PBF) Cardiac index (CI), ration of QP/QS. Right to left shunt will be quantified in liters per minutes as well as % of SBF and % of PBF.
  We will evaluate R-L shunt in normal conditions as well as after inducible Valsalva maneuver.
  Each patient will fill EQ-5D at the beginning of the study and Then 24 weeks after PFO closure.
Transesophageal Echocardiography examination before Patent foramen ovale closure | Up to 24 weeks (Prior subject's Patent foramen ovale closure)
  To evaluate the morphology of atrial septum
Evaluation of the severity of Right-Left shunt and comparison with atrial septal morphology | Up to 24 weeks
  Is there a significant correlation between atrial septal morphology and the level of severity of cardiac shunt as a predictive factor for systemic embolism
Spiroergometric examination with the measurement of VO2max | 6 months after Patent foramen ovale closure by means of a Patent foramen ovale occluder
  Detection of possible desaturation using the spiroergometric examination
Spiroergometric examination with the measurement of SpO2 | 6 months after Patent foramen ovale closure by means of a Patent foramen ovale occluder
  Detection of possible desaturation using the spiroergometric examination
Transesophageal Echocardiography routine examination after 6 months after Patent foramen ovale closure | Up to 24 weeks
  To evaluate results 6 months after Patent foramen ovale closure by means of a Patent foramen ovale occluder with a routine examination of Transesophageal Echocardiography
Influence of significant R-L shunt on exercise tolerance and quality of life of the patient | Up to 24 weeks
  To judge if the closure of Patent foramen ovale especially by the group of patients with significant R-L shunt may influence exercise tolerance and quality of patient life. Precise results of quantification of R-L Shunt will significantly correlated with a possible complications of PFO - systemic embolization, desaturation syndromes.

CONTACTS AND LOCATIONS:
Locations (6):
- Czechia (6):
  - Fakultní nemocnice Brno, Brno
  - I. interní kardioangiologická klinika, Fakultní nemocnice Hradec Králové, Hradec Králové
  - Fakultní nemocnice Ostrava, Ostrava
  - Všeobecná fakultní nemocnice v Praze, Prague
  - Institut klinické a experimentální medicíny (IKEM), Prague
  - Nemocnice Na Homolce, Prague

IPD SHARING:
Plan to Share IPD: No